CLINICAL TRIAL: NCT04038866
Title: Effects of Gait Rehabilitation With Dual Task in Patients With Parkinson's Disease: a Randomized Controlled Trial
Brief Title: Effects of Gait Rehabilitation With Dual Task in Patients With Parkinson's Disease
Acronym: DUALGAIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Asociación Parkinson Valencia (Other); Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Constanza San Martín, PhD Researcher at the Department of Medicine, Associate Professor at the Department of Physiotherapy, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT_DUALGAIT
Record Dates: First submitted 2019-07-25; First posted 2019-07-31 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Parkinson Disease
Keywords: gait biomechanics; physical rehabilitation; physical therapy; dual task
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Patients were randomized into two groups: control and experimental. Both groups performed different physical therapy programs to rehabilitate gait, in the experimental group they were included dual tasks during the walking exercises. Control and experimental group developed the rehabilitation programs at the same time.
Who Masked: Outcomes Assessor
Masking Description: The physiotherapists who assessment gait before and after interventions (post and follow-up) did not know to which group each patient belonged.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DUAL-TASK (Experimental): Patients with Parkinson's disease who carry out the rehabilitation gait with a dual-task program with secondary cognitive and upper limb motor tasks.
  In this group, the training of the tasks (walking and cognitive or motor) was performed separately and then they were trained at the same time under a progression system. Cognitive/motor secondary tasks were different from those used in the assessment of gait.
  Each training session consisted of three parts: the initial warm-up, dual-training, and back-to-calm.
  Interventions: Other: rehabilitation gait with dual task
- SINGLE-TASK (Active Comparator): Patients with Parkinson's disease who carry out the rehabilitation gait without a dual-task program (physical and walking exercises without additional load of cognitive or upper limb motor tasks).
  Each training session consisted of three parts: initial warm-up, physical exercise in single-task condition, and back-to-calm.
  The objectives and walking exercises were the same as those performed in the experimental group.
  Interventions: Other: rehabilitation gait without dual task

INTERVENTIONS:
Other: rehabilitation gait with dual task
  Arms: DUAL-TASK
Other: rehabilitation gait without dual task
  Arms: SINGLE-TASK

SUMMARY:
In functional environments, dual-tasks (DT) are common and require a correct motor and cognitive performance to be carried out successfully. In people with neurodegenerative diseases such as Parkinson's disease (PD), to walk with a secondary task affects gait. The inclusion of DT to the assessment and physical rehabilitation of patients allows to simulate day-to-day contexts in a controlled and safe environment and consequently, extrapolate more easily the advances of rehabilitation to daily life.

This project studied the effects of a gait rehabilitation program with dual tasks (DUALGAIT) in patients with Parkinson's disease and compared the results with a control active group of patients who performed a general physical rehabilitation program (without dual-task and only motor exercise practice).

The investigator's hypothesis is that gait training under dual conditions has a greater effect than traditional motor physiotherapy programs on the biomechanics of parkinsonian gait.

The present study is a randomized controlled clinical trial, with evaluators blind to the allocation of participants in the different groups.

DETAILED DESCRIPTION:
BACKGROUND AND OBJECTIVES

In functional environments, dual-tasks (DT) are common and require a correct motor and cognitive performance to be carried out successfully. In people with neurodegenerative diseases such as Parkinson's disease (PD), to walk with a secondary task affects gait causing an alteration of velocity, stride length, cadence and double support time and therefore, greater risk of falls. In fact, patients report gait impairments as the most disabling motor symptoms of the disease. The inclusion of DT to the assessment and physical rehabilitation of patients allows to simulate day-to-day contexts in a controlled and safe environment and consequently, extrapolate more easily the advances of rehabilitation to daily life. Advantages of this kind of training are not only functional, but it could induce neuroplasticity because it is a highly challenging activity for people with PD. While the neurophysiological changes of dual-task training are not yet known, the effects of training with dual-tasks on gait seem relatively clear. Studies so far have shown that improvements of spatiotemporal parameters of DT gait can be observed in integrated and consecutive DT training, which means that the addition of cognitive tasks into gait rehabilitation, either simultaneous or consecutively, is effective. However, there is not enough evidence that DT training is better than traditional EP training, i.e., including only motor training in single-task (ST) mode. The rest of the published studies include a passive control group (i.e. group that does not perform any type of control rehabilitation) or they correspond to repeated measures studies.

Additionally, there are other methodological issues that hinder the external validity of the experiments referenced so far. Firstly, the use of the same DT, both in training and evaluation of these effects training, could prevent to observe the transfers of these effects in untrained contexts. Secondly, the use of complex secondary tasks during the assessment such as mathematical tasks or recite alphabet letters may not be representative of the DT that occur in daily life. Thirdly, the different studies included the follow-up usually one month after the training, only one study evaluated the effects beyond this time. Finally, the lack of training done in a group, it prevents knowing if training with DT is possible in a group format, as well as individually at home.

Thus, this study aims:

1. To compare the short and mid-term effectiveness of a group dual-task program versus a group single-task program on biomechanics gait in people with PD.
2. To analyze the effect of dual-task therapy on clinical gait variables (standardized scales and tests), cognitive performance and quality of life.
3. To analyze the impact of secondary cognitive and motor tasks on single-gait before and after both physiotherapy programs.
4. To compare the parkinsonian gait before and after both therapies with normal gait from matched healthy subjects.

DESIGN

This was a single-blind, Randomized Control Trial (RCT) with 8-week follow-up and a convenience sample (specifically, modal instance sampling) in two parallel-group (experimental and active control group [1:1]) and one matched healthy control group and factorial design study.

BLINDING

Due to the nature of physical rehabilitation interventions, patients cannot be totally blind to the treatment that were performed and neither the treating physiotherapists, but the hypothesis and objectives of the study were hidden. At the same time, all participants were instructed to not divulge information regarding their intervention to the raters physiotherapists, who were blinded to group allocation in all assessment times. To control expectancy effects for patients it was explained that it is not yet determined which therapy is more effective. On the other hand, a code of consecutive numbers were assigned to the patients without pointing to the treatment group to which they belong.

RANDOMIZATION

The randomization process was performed by an extern researcher who is not involved in the development of the study. Stratified randomization will be performed by the severity stages of the disease (Hoehn & Yahr stages I, II and III) and participants were accordingly allocated to one of the two groups of physiotherapy treatment. Randomization was performed with a Microsoft Excel software with which a random sampling of half of the total of patients were extracted by the strata set for the dual-task program. After this, the treating physiotherapists will be responsible for the management and organization of the appointments of participants.

POWER CALCULATION

The sample size power calculation has been conducted based on the changes in the main outcomes of gait velocity evidenced in the literature in a verbal dual-task after a dual-gait training effect with PD patients. Previously, it has been shown that verbal tasks have great interference on Parkinsonian gait. For the sample size analysis, the Gpower software (Universität Kiel, Germany, Version 3.1) has been used [25]. A type I statistical error of 5% and a power of 80% was considered, which has resulted in 24 participants per group of treatment.

INTERVENTION

To ensure that the therapy sessions were carried out with a maximum of 10 people, the development of each program was repeated twice (DTP and STP), until completing the training of all recruited participants.

Both groups of the study (experimental and active comparator) performed 20 one-hour rehabilitation sessions, twice a week (10 weeks in total). All sessions of both groups were developed in a place provided by the researchers with the necessary elements for rehabilitation and in each of the sessions, there always were two physiotherapists. In each session, there were no more than ten patients.

1. Dual-task group Patients with Parkinson's disease carry out the rehabilitation gait with a dual-task program (DUALGAIT) with secondary cognitive and upper limb motor tasks.

   In this group, the training of walking and functional secondary tasks (cognitive or motor) first was separately (consecutive task training), to be performed later together in a dual-task (integrated dual-task training) with a progression system. Cognitive/motor secondary tasks were different from those used in the assessment of gait.

   Each training session consisted of three parts: the initial warm-up, dual-training, and back-to-calm.

   The objectives to walking improve and exercises were: i) Step/stride length with objective distance from 0.4 a 0.8 m in a progressive way and adapted to the heights of the participants, ii) Cadence/velocity training by digital metronome from 60 to 120 bpm, which in combination with the step lengths allowed the progressive training of walking velocity, iii) Lateral gait with lengths from 0.4 to 0.8 m., iv) Lower limb kinematics in support and swing phase through standardized practice of ankle, knee and hip movements during both phase, v) Arm swing practice during gait through elements, coordination with a partner and free, vi) Control of the flexor postural pattern by the practice of postural exercises and active movement that favor upright posture (neck extension, scapular adduction, shoulder retroversion, pelvic anteversion) and vii) Joint mobility and dissociation scapular-pelvic waist. In all of them, the use of external visual, auditory and verbal cues was included to provide the most objective feedback possible during motor learning.

   Additionally, the cognitive tasks used during the training were rehearsed in different positions (1st seated, 2nd biped and 3rd static gait) prior to the dual realization with the forward gait.

   The types of secondary tasks trained were: 1) verbal fluency, 2) auditory recognition, 3) visual recognition, 4) mathematical calculation, 5) memory, 6) visuospatial planning, 7) fine motor skills, 8) motor task of money manipulation, 9) motor transport task and 10) motor task of transferring an object to another person. Each task category had a level of complexity (basic, medium and high).
2. Single-task group Patients with Parkinson's disease carry out the rehabilitation gait without a dual-task program (physical and walking exercises without an additional load of cognitive or upper limb motor tasks). Each training session consisted of three parts: initial warm-up, physical exercise in single-task condition, and back-to-calm. The objectives and walking exercises were the same as those performed in the experimental group.

SUBJECTS

Forty participants completed the study, 23 performed the dual-task physiotherapy program and composed the Dual-task group (DTG), while the other 17 formed the Single-task group (STG). All patients came from the La Fe Clinical and Polytechnic Hospital (Valencia, Spain) completed all phases of the study. The patients were recruited with the diagnosis made by a neurological doctor. All participants signed informed consent prior to their participation in the study, then they were randomly assigned to one of the rehabilitation groups (DTG and STG).

TEST PROCEDURE

Before conducting the biomechanics gait assessments, a previous evaluation was carried out to verify the eligibility criteria. This valuation session was held a few days before the biomechanics gait assessment prior to the intervention and the following was verified:

* Registration of sociodemographic data and neurological history
* Anthropometric evaluation
* Clinical evaluation of Parkinson's disease (Disease duration, Hemibody where signs predominate, Hoehn & Yahr stage, New Freezing of Gait Questionnaire)
* Cognitive state (Mini-mental test adapted for Parkinson's disease).

After determining the eligibility criteria, three assessments sessions were carried out at the University of Valencia laboratories. These were: 1) immediately before starting the rehabilitation program (Baseline), 2) immediately after completing the rehabilitation program (Postintervention) and 3) eight weeks after completing the rehabilitation program (8-week follow-up). Between Postintervention and 8-week follow-up tests, participants did not perform any kind of physical therapy, sports or physical activity. Participants were evaluated in the on-medication state. In each of the assessment sessions biomechanics of gait, the clinical performance of mobility, balance and gait, and cognition were evaluated.

The biomechanics gait evaluation was carried out in a corridor 10m long and data were registered using 3D photogrammetry with 12 smart cams (Kinescan/IBV software, Biomechanical Institute of Valencia, Valencia, Spain, version 5.3.0.1) and two force platforms (Dinascan/IBV Biomechanical Institute of Valencia, Valencia, Spain). All the participants walked at a self-selected comfortable speed, barefoot and under five conditions: i) single task (ST): walking without secondary tasks with the attention focused only on walking performance, ii) visual dual-task (viDT): walking while watching the time on an analog clock projected at the end of the walkway, iii) verbal dual-task (veDT): walking while telling the evaluator the activities they had performed the previous day in a chronological order, iv) auditory dual-task (aDT): walking while listening and recognizing different daily noises and, v) motor dual-task (mDT): walking while carrying one glass in each hand and repeatedly transferring their contents from one to the other. During DT gait, participants were urged to focus attention on the secondary task. For each of the five evaluated walking conditions, 10 repetitions were performed, five with each foot, to later use their average. Before recording gait, participants were allowed to walk in the corridor (ST condition) to familiarize themselves with the test.

The biomechanics outcomes were:

1. Spatio-temporal outcomes: velocity (m/s), stride length (m), cadence (steps/min), double support time (% of gait cycle) and step width (m).
2. kinematics outcomes: range of motion of the ankle (°), maximum hip extension (°), maximum hip flexion (°).
3. Kinetic outcomes: vertical reaction force 1 (N), vertical reaction force 2 (N), anterior-posterior reaction force 1 (N).

On the other hand, to know if the effects of the treatments would be detectable with the clinical tests and scales, a Dynamic Parkinson Gait Scale (DYPAGS), Tinetti Mobility Test, both total score (TinettiT) and scores from subtest gait (TinettiG) and balance (TinettiB) and Time up and go test (TUG) were used. Finally, we used the Trail making test, parts A (TMTa) and B (TMTb) to evaluate executive cognitive performance and the Parkinson's disease questionnaire-39 (PDQ-39) for quality of life assessment.

STATISTIC ANALYSIS

Statistical analyses were performed using SPSS v.24 (SPSS Inc., Chicago, IL, USA). Mean and standard deviations (SD) were calculated. A three-factor mixed Multivariate Analysis of Variance (MANOVA) was conducted to analyze their effects on the biomechanical dependent variables previously described in table 3. The within-subject factors are rehabilitation with three categories (Baseline, Postintervention and Follow-up) and conditions, with five categories (ST, viDT, veDT, aDT and mDT). The between-subject factor is group with two categories (DTG and STG). Stride length was standardized by the lower limb length of participants. In addition, a two-factor mixed MANOVA was conducted to analyze the effects of within-subject factors rehabilitation and the between-subject factor group on the clinical tests. When significant effects are found, Bonferroni was used for post hoc comparisons. Differences was declared statistically significant if p<0.05.

To check for differences between the demographic outcomes between groups, multivariate one-way analysis with the between-subject factor group was conducted. Furthermore, to test for sex differences between groups, a chi-square test was used.

Before the statistical analysis, the following assumptions were checked: 1) Normality, the distribution of the residuals was tested using the Shapiro-wilk test, 2) Sphericity, the homogeneity between variances of the differences between pairs of measures was checked with the Mauchly sphericity test, 3) Homoscedasticity, homogeneity of variances was evaluated using the Levene test, 4) Equality of covariance matrices, the equality of variance-covariance matrices across the cells formed by the between-subjects effects was tested with the Box's M test, 5) Absence of multicollinearity, the correlation level between dependent variables were observed with the Pearson correlation test. When any of these assumptions were not met, the necessary statistical corrections were used.

TIMING OF THE STUDY

* Resolution Ethics Committee of the University of Valencia (Spain): May 14, 2014.
* Resolution Ethics Committee of the Biomedical Research of La Fe University and Polytechnic Hospital (Valencia, Spain): September 9, 2014.
* Start of recruitment of participants: June 14, 2014.
* Completion of participant evaluations: June 30, 2016.
* Data pretreatment, statistical analysis and dissemination of results: from september 2016 to present.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD
* To present Hoehn & Yahr stadium (H & Y) I, II or III
* Minimum of two months without any kind of physical rehabilitation.
* To be able to walk by themselves,
* To have a normal cognitive state according to the Minimental test adapted for PD
* Symmetry in lower limb length (<1cm).

Exclusion Criteria:

* Presence of another symptomatic neurological or musculoskeletal disease
* History of trauma or surgery on the lower limbs
* Balance disorders due to other diseases
* Uncontrolled chronic diseases (e.g. hypertension or diabetes).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-06-14 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Velocity | 20 weeks (time that includes 10 weeks of training, 8 weeks of follow-up and one week before and after the entire study to perform the Basal and Follow-up measurements)
  distance travelled by the body per unit of time (m·s-1)

SECONDARY OUTCOMES:
Stride length | 20 weeks
  distance measured between two consecutive heel strikes of the same foot (m)
Cadence | 20 weeks
  number of steps taken in a minute (steps·min-1)
Double support time | 20 weeks
  sum of the amount of time in which there is double-limb support in a walking cycle (%)
range of motion of the ankle | 20 weeks
  sum of maximum angle of plantar flexion and maximum angle of dorsiflexion of the foot (°)
Maximum hip extension | 20 weeks
  maximum extension angle reached by the hip joint during the stance phase of the gait cycle (°)
Maximum hip flexion | 20 weeks
  maximum flexion angle reached by the hip joint during the swing phase of the gait cycle (°)
Vertical reaction force 1 | 20 weeks
  milestone of the vertical component curve of reaction forces corresponding to the heel strike of the gait cycle
Vertical reaction force 2 | 20 weeks
  milestone of the vertical component curve of reaction forces corresponding to the mid stance of the gait cycle (N)
Anterior-posterior reaction force 1 | 20 weeks
  milestone of anteroposterior component curve of reaction force that corresponds to the braking impulse

CONTACTS AND LOCATIONS:
Overall Officials: Constanza I San Martín Valenzuela, PhD, Principal Investigator — Faculty of Medicine, University of Valencia; Pilar Serra Añó, PhD, Study Director — Faculty of Physiotherapy, University of Valencia; José Manuel Tomás Miguel, PhD, Study Director — Faculty of Psychology, University of Valencia
Locations (1):
- University of Valencia, Faculty of Medicine, Unit of evaluation in personal autonomy, dependence and mental disorders, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
All the information of the study, as well as its results, will be shared in scientific publications and conferences related to the research area.
  The information that is intended to be published in scientific journals includes: 1) Study Protocol, 2) Statistical Analysis, 3) Informed Consent Form, 4) Clinical Study Results.

REFERENCES:
- [Background] Strouwen C, Molenaar EA, Keus SH, Munks L, Munneke M, Vandenberghe W, Bloem BR, Nieuwboer A. Protocol for a randomized comparison of integrated versus consecutive dual task practice in Parkinson's disease: the DUALITY trial. BMC Neurol. 2014 Mar 27;14:61. doi: 10.1186/1471-2377-14-61. PMID 24674594
- [Background] Brauer SG, Woollacott MH, Lamont R, Clewett S, O'Sullivan J, Silburn P, Mellick GD, Morris ME. Single and dual task gait training in people with Parkinson's disease: a protocol for a randomised controlled trial. BMC Neurol. 2011 Jul 27;11:90. doi: 10.1186/1471-2377-11-90. PMID 21791117
- [Result] Geroin C, Nonnekes J, de Vries NM, Strouwen C, Smania N, Tinazzi M, Nieuwboer A, Bloem BR. Does dual-task training improve spatiotemporal gait parameters in Parkinson's disease? Parkinsonism Relat Disord. 2018 Oct;55:86-91. doi: 10.1016/j.parkreldis.2018.05.018. Epub 2018 May 18. PMID 29802080
- [Result] Strouwen C, Molenaar EALM, Munks L, Broeder S, Ginis P, Bloem BR, Nieuwboer A, Heremans E. Determinants of Dual-Task Training Effect Size in Parkinson Disease: Who Will Benefit Most? J Neurol Phys Ther. 2019 Jan;43(1):3-11. doi: 10.1097/NPT.0000000000000247. PMID 30531381
- [Result] Strouwen C, Molenaar EALM, Munks L, Keus SHJ, Zijlmans JCM, Vandenberghe W, Bloem BR, Nieuwboer A. Training dual tasks together or apart in Parkinson's disease: Results from the DUALITY trial. Mov Disord. 2017 Aug;32(8):1201-1210. doi: 10.1002/mds.27014. Epub 2017 Apr 25. PMID 28440888
- [Result] Fok P, Farrell M, McMeeken J. The effect of dividing attention between walking and auxiliary tasks in people with Parkinson's disease. Hum Mov Sci. 2012 Feb;31(1):236-46. doi: 10.1016/j.humov.2011.05.002. Epub 2011 Jul 1. PMID 21723639
- [Result] Fok P, Farrell M, McMeeken J. Prioritizing gait in dual-task conditions in people with Parkinson's. Hum Mov Sci. 2010 Oct;29(5):831-42. doi: 10.1016/j.humov.2010.06.005. Epub 2010 Aug 19. PMID 20727609
- [Result] Yogev-Seligmann G, Giladi N, Brozgol M, Hausdorff JM. A training program to improve gait while dual tasking in patients with Parkinson's disease: a pilot study. Arch Phys Med Rehabil. 2012 Jan;93(1):176-81. doi: 10.1016/j.apmr.2011.06.005. Epub 2011 Aug 17. PMID 21849167
- [Result] Mirelman A, Maidan I, Herman T, Deutsch JE, Giladi N, Hausdorff JM. Virtual reality for gait training: can it induce motor learning to enhance complex walking and reduce fall risk in patients with Parkinson's disease? J Gerontol A Biol Sci Med Sci. 2011 Feb;66(2):234-40. doi: 10.1093/gerona/glq201. Epub 2010 Nov 24. PMID 21106702
- [Result] Brauer SG, Morris ME. Can people with Parkinson's disease improve dual tasking when walking? Gait Posture. 2010 Feb;31(2):229-33. doi: 10.1016/j.gaitpost.2009.10.011. Epub 2009 Dec 6. PMID 19969461
- [Result] Canning CG, Ada L, Woodhouse E. Multiple-task walking training in people with mild to moderate Parkinson's disease: a pilot study. Clin Rehabil. 2008 Mar;22(3):226-33. doi: 10.1177/0269215507082341. PMID 18285432
- [Derived] San Martin Valenzuela C, Moscardo LD, Lopez-Pascual J, Serra-Ano P, Tomas JM. Effects of Dual-Task Group Training on Gait, Cognitive Executive Function, and Quality of Life in People With Parkinson Disease: Results of Randomized Controlled DUALGAIT Trial. Arch Phys Med Rehabil. 2020 Nov;101(11):1849-1856.e1. doi: 10.1016/j.apmr.2020.07.008. Epub 2020 Aug 12. PMID 32795562
- [Derived] San Martin Valenzuela C, Duenas Moscardo L, Lopez-Pascual J, Serra-Ano P, Tomas JM. Interference of functional dual-tasks on gait in untrained people with Parkinson's disease and healthy controls: a cross-sectional study. BMC Musculoskelet Disord. 2020 Jun 22;21(1):396. doi: 10.1186/s12891-020-03431-x. PMID 32571284